CLINICAL TRIAL: NCT01669187
Title: Phase 1 of the The Effects of Pre-operative Physical Therapy Education and Exercise on Patient Outcomes Post Breast Cancer Surgery: a Randomized Controlled Trial
Brief Title: The Effects of Pre-operative Physical Therapy Education
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study withdrawn.
Sponsor: Oakland University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OU-4824
Record Dates: First submitted 2012-07-20; First posted 2012-08-20 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education brochure (Active Comparator): The control group will receive a standard education brochure which will be provided pre-operatively to the participants.
  Interventions: Other: Education brochure
- Live education and exercise instruction (Experimental): The intervention group will receive one to two physical therapy visits consisting of education on the lymphedema risks and prevention factors, along with detailed information about what to except post-surgery as well as with radiation/chemotherapy. Additionally, those in the intervention group will be instructed on exercises to maintain or increase glenohumeral and scapulothoracic joint ROM post surgery and will be set up with a walking program.
  Interventions: Other: Live education and exercise instruction

INTERVENTIONS:
Other: Education brochure
  Arms: Education brochure
Other: Live education and exercise instruction — Participants will receive one to two physical therapy visits consisting of education on the lymphedema risks and prevention factors, along with detailed information about what to except post-surgery as well as with radiation/chemotherapy. Additionally, those in the intervention group will be instructed on exercises to maintain or increase glenohumeral and scapulothoracic joint ROM post surgery and will be set up with a walking program.
  Arms: Live education and exercise instruction

SUMMARY:
It is expected that patients who receive physical therapy before surgery will have greater range of motion (ROM), strength, function, satisfaction, and less swelling, pain, and anxiety following surgery compared to those in the control group.

ELIGIBILITY:
Inclusion Criteria:

* be over the age of 18,
* have a good understanding of the English language, and
* be scheduled to undergo either a mastectomy, lumpectomy, ALND or Sentinel Lymph Node Dissection (SLND) with or without breast reconstruction.

Exclusion Criteria:

* if they previously underwent one of the previously mentioned procedures mastectomy, lumpectomy, ALND or Sentinel Lymph Node Dissection (SLND) with or without breast reconstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in score for Shoulder Pain and Disability Index (SPADI) | Before sugery (range 0-4 weeks before surgery), 2 weeks post operatively and 6 weeks post-operatively
  Functional outcome measure questionnaire

SECONDARY OUTCOMES:
Change in Shoulder range of motion with goniometer | Pre-operatively (0-4 weeks pre-operatively), 2 and 6 weeks post-operatively

OTHER OUTCOMES:
Change in other physical therapy test and measures | Once pre-operatively (0-4 weeks before surgery), 2 and 6 weeks after surgery
  6 minute walk test; presence of cording; number of patient reported medical complications; shoulder strength measured by a dynamometer; Arm lymphedema measured by volumeter; Anxiety, general functional abilities, and QOL will be measured by the Functional Assessment of Cancer Therapy- Breast Cancer (FACT-B); Patient satisfaction will be measured using a 5 point Likert Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Eve S Pepin, DPT, Principal Investigator — Oakland University
Locations (2):
- United States (2):
  - St-Mary's of Michigan, Saginaw, Michigan
  - St. Mary's of Michigan, Saginaw, Michigan